CLINICAL TRIAL: NCT04403308
Title: An Open-label, Uncontrolled, Dose Escalation Study in Patients With Advanced or Metastatic Solid Cancers (ONO-7913-01)
Brief Title: ONO-7913 Phase I Study (ONO-7913)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONO-7913-01
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ONO-7913 as a Single Agent (Experimental)
  Interventions: Biological: ONO-7913

INTERVENTIONS:
Biological: ONO-7913 — ONO-7913 will be administered by intravenous continuous infusion during the designated time.

SUMMARY:
To assess the tolerability, safety, and pharmacokinetics (PK) of ONO-7913 in patients with advanced or metastatic solid cancers and explore its efficacy and biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed advanced or metastatic solid tumors
2. ECOG Performance Status of 0-1
3. Patients with life expectancy of at least 3 months

Exclusion Criteria:

1. Patients with multiple cancers
2. Patients with history of serious allergy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-01-13 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities | 28 days
  Number of participants with a DLT
Adverse events | Up to 24 months
  Assessed by the NCI CTCAE v5.0 criteria

SECONDARY OUTCOMES:
Concentration vs time of ONO-7913 as single dose | Up to 24 months
  PK profile

CONTACTS AND LOCATIONS:
Overall Officials: Kazuhiro Nakabayashi, Study Chair — Ono Pharmaceutical Co. Ltd
Locations (1):
- Local Institution, Chuo-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No